CLINICAL TRIAL: NCT01908088
Title: Autologous Transplantation of Cultured Fibroblast on Amniotic Membrane for Mitten Hand Deformity in Patients With Epidermolysis Bullosa
Brief Title: Autologous Transplantation of Cultured Fibroblast on Amniotic Membrane in Patients With Epidermolysis Bullosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Collaborators: Hazrat Fatemeh Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-skin-003
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2010-02

CONDITIONS: Epidermolysis Bullosa With Mitten Hands
Keywords: Epidermolysis Bullosa mitten hand deformity autologous cultured fibroblast; amniotic membrane
MeSH Terms: interventions — Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fibroblast transplant (Experimental): Transplantation of autologous cultured fibroblast on amniotic membrane in patients with Epidermolysis Bullosa with mitten hand deformity
  Interventions: Biological: Cell transplantation

INTERVENTIONS:
Biological: Cell transplantation — autologous transplantation of cultured fibroblast on amniotic membrane in patients with Epidermolysis Bullosa with mitten hands.
  Other Names: autologous transplantation of cultured fibroblast on amniotic membrane

SUMMARY:
Epidermolysis Bullosa (EB) is a blistering disease that is caused by defective anchoring fibrils and hemidesmosome in basement membrane of the skin layer. EB is inherited either autosomal or recessive and has 3 types. Recessive Dystrophic Epidermolysis Bullosa (RDEB) is severe with some morbidity such as mitten hand deformity.

The management of these patients is very difficult because no effective treatment has been known yet.

The EB patients with mitten hand deformity need surgery to have a biologic dressing for areas of hand which is without the skin. In this study the investigators assess the safety of autologous transplantation of cultured fibroblast on amniotic membrane (AM,as coverage) for them.

DETAILED DESCRIPTION:
Epidermolysis Bullosa patients with mitten hand deformity were included. (based on inclusion & exclusion criteria) These patients should be offered for surgery to release the adhesions between fingers and MCP. When the consent form was accepted and the lab test was confirmed, a small skin biopsy was removed from retro auricle and fibroblast cells were separated and cultured. These cells were seeded on AM and the microbial test was done as evidence to prove the safety.

Under general anesthesia, when the hands adhesion was removed, the autologous fibroblast cultured on AM was transplanted to the both hands (specially the area without skin coverage) and the hands were dressed afterward.

The dressing was changed and the wound was checked regularly to detect any complications.

ELIGIBILITY:
Inclusion Criteria:

* Both genders Age: 5-25y No history of other systemic disease No history of other cell therapy method No infection in donor or recipient site HCV Ab/HIV Ab/ HBS Ag tests were negative

Exclusion Criteria:

* Age less than 5y or more than 25y. History of other systemic disease History of other cell therapy method Infection in donor or recipient site Positive Lab tests for contagious viral diseases Pregnancy or lactating History of malignancy

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain | 1month
  Evaluation the pain reduction 1 month after cell transplantation by VAS scoring.
Infection | 1week
  Evaluation the symptoms of any infection in the site of transplantation during 1week after transplantation.
Bleeding | 1week
  Evaluation the presence of any bleeding at the site of transplantation during 1 week after transplantation.
Healing | 1month
  Evaluation the healing of ulcers 1month after transplantation base on changing the dressing time.

SECONDARY OUTCOMES:
new ulceration | 3months
  Evaluation the new blister or ulceration during 3 to 6 months after transplantation.
Range of motion | 6months
  Evaluation the range of hand motion between 0 -110 for every fingers 6 months after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan Institute Cell Therapy Center; Saeed Shafiyan, MD, Study Director — Dermatogist,Depatment of Regenerative medicin of Royan Institute; Zahra Orouji, MD, Principal Investigator — Regenerative Medicine Department of Royan Institute; Kamal Seyed Forootan, MD, Principal Investigator — Plastic Surgoen, Hazrat Fatemeh Hospital; Seyed Mohammad Javad Fatemi, MD, Principal Investigator — Plastic Surgoen,Hazrat Fatemeh Hospital
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.org